CLINICAL TRIAL: NCT01026337
Title: An Imaging and Histopathologic Study to Predict Response to Sunitinib Therapy in Patients With Metastatic or Locally Advanced Renal Cell Carcinoma
Brief Title: Magnetic Resonance Imaging (MRI) in Predicting Response to Sunitinib Malate in Patients With Locally Advanced or Metastatic Kidney Cancer
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 03809; NCI-2009-01414; NCT00915993 (obsolete NCT alias)
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Renal Cell Carcinoma; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer
Keywords: recurrent renal cell cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib; Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arm I: Patients receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 42 days in the absence of disease progression or unacceptable toxicity.
  Patients undergo dynamic contrast-enhanced MRI at baseline and after the first 4 weeks of sunitinib malate.
  Interventions: Genetic: mutation analysis; Other: pharmacological study; Procedure: dynamic contrast-enhanced magnetic resonance imaging; Drug: sunitinib malate; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: mutation analysis — Correlative study
Other: pharmacological study — Correlative study
  Other Names: pharmacological studies
Procedure: dynamic contrast-enhanced magnetic resonance imaging — Undergo DCE-MRI
  Other Names: DCE-MRI
Drug: sunitinib malate — Given orally
  Other Names: SU011248; SU11248; sunitinib; Sutent
Other: immunohistochemistry staining method — Correlative study
  Other Names: immunohistochemistry
Other: laboratory biomarker analysis — Correlative study

SUMMARY:
Rationale: Diagnostic procedures, such as MRI, may help doctors predict a patient's response to treatment and help plan the best treatment.

Purpose: This clinical trial is studying MRI in predicting response to sunitinib malate in patients with locally advanced or metastatic kidney cancer.

DETAILED DESCRIPTION:
Primary Objectives:

I. To correlate tumor vascular permeability by DCE-MRI with clinical outcome for patients treated with sunitinib (PFS).

II. To correlate genetic and histologic characteristics of the primary tumor with vascular permeability by DCE-MRI.

Secondary Objectives:

I. To correlate genetic and histologic characteristics of the primary tumor with clinical outcome for patients treated with sunitinib.

II. Samples will be collected for potential future exploratory analyses of pharmacokinetic and pharmacogenomic parameters.

Outline: Patients receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 42 days in the absence of disease progression or unacceptable toxicity.

Patients undergo dynamic contrast-enhanced MRI at baseline and after the first 4 weeks of sunitinib malate.

ELIGIBILITY:
Inclusion

* AJCC stage IV or locally advanced (or inoperable) renal cell carcinoma for which archival tissue is available
* No prior anti-angiogenic therapy
* Prior radiation therapy to a symptomatic site of disease is allowed
* ECOG performance status of 0, 1 or 2
* White Blood Count >= 3,000/mm^3
* Absolute Granulocyte Count >= 1,500/mm^3
* Platelet Count >= 100,000/mm^3
* Serum creatinine =< 2.0 x upper limit of normal (ULN) OR serum creatinine clearance (CrCl) >= 40 ml/min
* Total Bilirubin =< 1.5 x ULN (< 3.0 x ULN in the presence of Gilbert's disease)
* AST/ALT =< 2.5 x ULN (=< 5.0 ULN in the presence of liver metastases)
* INR =< 1.5 and a PTT within normal limits; patients who are taking warfarin must have documentation of an INR =< 1.5 and a PTT within normal limits prior to the initiation of anticoagulation to rule out a baseline coagulopathy
* Patient must not have pre-existing thyroid abnormality with thyroid stimulating hormone that cannot be maintained in the normal range with medication
* Patient must not have hypertension that cannot be controlled by medications (diastolic blood pressure >= 100 mm Hg despite optimal medical therapy)
* Patient must not have ongoing cardiac dysrhythmias of NCI CTCAE Version 3.0 grade >= 2
* Patients must not receive any other investigational agents during the period on study
* Patients must not have a history or clinical evidence of brain metastasis; however, patients with resected or radiated brain metastases are eligible
* Patients must not have a serious intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics, clinically significant cardiovascular disease (e.g., uncontrolled hypertension, myocardial infarction, unstable angina), New York heart association grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication
* Patients must not have a serious intercurrent illness including, but not limited to, grade II or greater peripheral vascular disease within 1 year prior to study entry, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not be taking cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine or phenobarbital), rifampin or St. John's wort
* Women must not be pregnant or breast-feeding
* All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal, barrier method of birth control, or abstinence) prior to study entry and for the duration of study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-04; Primary Completion 2015-12 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Progression-free survival
Correlation of tumor vascular permeability as measured by dynamic contrast-enhanced MRI with clinical outcome and with tumor angiogenesis as measured by immunohistochemistry (IHC)

SECONDARY OUTCOMES:
Tumor regression as measured by Response Evaluation Criteria In Solid Tumors (RECIST) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Keefe, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States